CLINICAL TRIAL: NCT01563497
Title: A Phase 1, Open-Label, Single Dose, Bioavailability Study In Healthy Volunteers Comparing PF-05089771 TS Tablet To PF-05089771 TS Oral Dispersion In The Fasted State And To PF-05089771 TS Tablet In The Fasted And The Fed State
Brief Title: A Study Comparing PF-05089771 TS Tablet to PF-05089771 TS Oral Dispersion In The Fasted State And To PF-05089771 TS Tablet In The Fasted And Fed State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B3291007
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — PF-05089771

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-05089771 Oral Dispersion fasted (Experimental): Oral dispersion TS formulation- fasted
  Interventions: Drug: PF-05089771
- PF-05089771 TS formulation fasted (Experimental): Tablets TS formulation- fasted
  Interventions: Drug: PF-05089771
- PF-05089771 TS formulation fed (Experimental): Tablets TS formulation- fed
  Interventions: Drug: PF-05089771

INTERVENTIONS:
Drug: PF-05089771 — Oral dispersion TS formulation- fasted
  Arms: PF-05089771 Oral Dispersion fasted
Drug: PF-05089771 — Tablets TS formulation- fasted
  Arms: PF-05089771 TS formulation fasted
Drug: PF-05089771 — Tablets TS formulation- fed
  Arms: PF-05089771 TS formulation fed

SUMMARY:
The primary purpose of this study is to estimate the relative bioavailability and food effect of a PF-05089771 tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or non-childbearing potential female subjects between the ages of 18 and 55 years

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal,endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug within 60 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* Screening supine blood pressure ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), on a single measurement (confirmed by a single repeat, if necessary) following at least 5 minutes of rest 7. Single 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 mseca at screening. If QTc exceeds 450 msec, or QRS exceeds >120 mseca the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) for PF-05089771 in plasma (measured in ng/mL) | days 1-3
AUClast = Area under the curve from the time of dosing to the last data point taken (ng.hr/mL) | days 1-3
AUCinf = Area under the curve from the time of dosing extrapolated to infinity (ng.hr/mL) | days 1-3
Tmax = Time of maximum concentration of PF-05089771 in plasma (hr) | days 1-3
t½ = Elimination half life of PF-05089771 (hr) | days 1-3

SECONDARY OUTCOMES:
evaluation of safety clinical laboratory tests, vital signs, ECGs, physical examinations and adverse event monitoring. | days 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3291007&StudyName=A%20Study%20Comparing%20PF-05089771%20TS%20Tablet%20to%20PF-05089771%20TS%20Oral%20Dispersion%20In%20The%20Fasted%20State%20And%20To%20PF-05089771%20TS%20Tablet%20In%20The%20